CLINICAL TRIAL: NCT05351203
Title: Ultrasound Guide Bilateral Erector Spinae Block Versus Caudal Epidural Analgesia for Perioperative Analgesia in Lumbar Spine Surgeries:Randomized Controlled Study
Brief Title: Ultrasound Guided Bilateral Erector Spinae Block Versus Caudal in Lumbar Spine Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abd elmoneim Adel Abd elmoneim, clinical professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MS-620-2021
Record Dates: First submitted 2022-04-18; First posted 2022-04-28 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Acute Postoperative Pain
Keywords: caudal; Erector spinae block; lumbar surgery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- caudal epidural group (Active Comparator): the patient will be positioned in prone position, sterilized from the iliac crest margin to the lower buttock by betadine three times and will be covered by sterile drapes exposing the sacral area. Sacral horns will be palpated and sacral hiatus and epidural area will be determined at S4-S5 level through the ultrasound linear transducer probe that is covered in sterile plastic bag . Short axis (transverse) is used first to identify the two sacral cornua as two hyperechoic reverse U-shaped structure "Frog sign" and the sacrococcygeal ligament in between and epidural space beneath. An 18-gauge epidural needle (length 90 mm) is used for direct puncture of sacrococcygeal membrane out of plane then the probe is rotated to long axis (longitudinal) and the needle is seen in plane in the epidural space. Injection of 30 ml 0.125% bupivacaine will expand the epidural space.
  Interventions: Procedure: caudal block
- Erector spinae group (Experimental): ● The patient will be in the prone position, after skin sterilization, ESP block will be performed at the level of L3. a curvilinear high-frequency ultrasound transducer (Siemens acuson x300 3-5 MHz ultrasound) will be placed sagittal 3 cm lateral to L3 spinous process where a hyperechoic shadow of the transverse process (TP) and erector spinae will be defined. A 22-gauge spinal needle will be inserted in cranial to caudal direction toward TP in plane to the ultrasound transducer until the needle touches the TP crossing the whole muscles. The location of the needle tip will be confirmed by visible normal saline solution separating erector spinae muscle off the bony shadow of the TP on ultrasound imaging. After confirming the needle site, 30 mL of 0.25% bupivacaine will be injected. The procedure will be repeated following the same steps on the other side.
  Interventions: Procedure: Erector spinae block

INTERVENTIONS:
Procedure: caudal block — . Sacral horns will be palpated and sacral hiatus and epidural area will be determined at S4-S5 level through the ultrasound,. Short axis (transverse) is used first to identify the two sacral cornua as two hyperechoic reverse U-shaped structure "Frog sign" and the sacrococcygeal ligament in between and epidural space beneath. An 18-gauge epidural needle (length 90 mm) is used for direct puncture of sacrococcygeal membrane out of plane then the probe is rotated to long axis (longitudinal) and the needle is seen in plane in the epidural space. Injection of 30 ml 0.125% bupivacaine will expand the epidural space.
  Other Names: caudal epidural block
  Arms: caudal epidural group
Procedure: Erector spinae block — ● The patient will be in the prone position, after skin sterilization, ESP block will be performed at the level of L3. a curvilinear high-frequency ultrasound transducer (Siemens acuson x300 3-5 MHz ultrasound) will be placed sagittal 3 cm lateral to L3 spinous process where a hyperechoic shadow of the transverse process (TP) and erector spinae will be defined. A 22-gauge spinal needle will be inserted in cranial to caudal direction toward TP in plane to the ultrasound transducer until the needle touches the TP crossing the whole muscles. The location of the needle tip will be confirmed by visible normal saline solution separating erector spinae muscle off the bony shadow of the TP on ultrasound imaging. After confirming the needle site, 30 mL of 0.25% bupivacaine will be injected. The procedure will be repeated following the same steps on the other side.
  Other Names: ESP block
  Arms: Erector spinae group

SUMMARY:
Major lumbar spine surgeries are associated with severe postoperative pain that usually lasts for at least 3 days.Caudal epidural analgesia has a crucial role in providing effective pain relief post lumbar spine surgeries by blocking sensory input at the level of the spinal cord. Erector Spinae Plane Block (ESPB) as a new technique of trunk fascia block was proposed in 2016Reports showed that ESPB significantly relieved postoperative pain in patients with lumbosacral spine surgery, reducing the use of analgesics.

The aim of this work is to evaluate the pre-emptive analgesic effect of Ultrasound guided bilateral erector spinae block Vs Caudal epidural analgesia in Lumbar spine surgeries during peri-operative period.

Objectives:

* To assess the duration of analgesia in both groups and time to rescue analgesia .
* To assess Visual analogue scale (VAS) score in both groups.
* To assess complications of both groups

DETAILED DESCRIPTION:
This is a randomized controlled study designed to include 50 patients aged from 18 to 65 years old undergoing lumbar spine surgeries.

fifty patients meeting the inclusion criteria will be randomly assigned into two equal groups: Group A(n=25): caudal epidural group. Group B(n=25): bilateral ultrasound guided Erector spinae block group.

All patients will be assessed clinically and investigated for exclusion of any of the above mentioned contraindications. Laboratory work needed will be: Complete blood count (CBC); prothrombin time and concentration (PT& PC); partial thromboplastin time (PTT); bleeding time (BT); clotting time (CT) , liver function tests and kidney function tests .

● Operating Room preparation & Equipment: The ultrasound used will be SonoSite M Turbo (USA), the scanning probe will be the linear multi-frequency 6-13 megahertz transducer (L25 x 6-13 MHz linear array).

Methods:

General anaesthesia will be induced. 1.5 μg/kg fentanyl based on lean body weight with maximum dose of 200 μg and 2 mg/kg propofol will be given based on total body weight. (14) Tracheal intubation will be facilitated with 0.5 mg/kg atracurium based on ideal body weight. (15) . The surgical intervention will be then allowed 20 minutes after finishing the block procedure.

Volume controlled ventilation will be adjusted to maintain normocapnia. Anesthesia will be maintained by using 1.5% isoflurane in a mixture of oxygen and air (50/50) and atracurium top ups at a dose of 0.1mg/kg every 30 minutes.

Patients will be placed in the prone position on a Relton Hall frame or padded bolsters.

All participants will be given 1 gram of intravenous paracetamol with maximum dose of 4 gm every 24 hour, together with 4 mg ondansetron 10 min prior to the end of surgery for postoperative nausea and vomiting prophylaxis.

Failed block (increase in Heart rate (HR) and mean arterial blood pressure (MABP)>20% from base line with skin incision) will be treated by 1 ug/kg of fentanyl as top-up doses and increasing isoflurane concentration in case of inadequate response to fentanyl.

After skin closure, inhalational anesthesia will be discontinued and reversal of muscle relaxation with atropine (0.02 mg/Kg) and neostigmine (0.05 mg/Kg) will be administered intravenous after return of patient's spontaneous breathing. Patients will then be transferred to post anesthesia care unit (PACU) for 60 min to complete recovery and monitoring.

* At any time hypotension (defined as a decrease in mean arterial pressure (MAP) >25% from baseline value or systolic arterial pressure (SAP <100 mmHg)) will be treated with 5 mg IV bolus ephedrine and repeated every 3 minutes until the hypotension resolved. Bradycardia (defined as a HR <40 beats per minute) will be treated with atropine 0.5 mg IV.
* In group (A): Caudal Epidural Analgesia
* For the caudal block, the patient will be positioned in prone position, sterilized from the iliac crest margin to the lower buttock by betadine three times and will be covered by sterile drapes exposing the sacral area. Sacral horns will be palpated and sacral hiatus and epidural area will be determined at S4-S5 level through the ultrasound transducer that is covered in sterile plastic bag . Short axis (transverse) is used first to identify the two sacral cornua as two hyperechoic reverse U-shaped structure "Frog sign" and the sacrococcygeal ligament in between and epidural space beneath. An 18-gauge epidural needle (length 90 mm) is used for direct puncture of sacrococcygeal membrane out of plane then the probe is rotated to long axis (longitudinal) and the needle is seen in plane in the epidural space. Injection of 30 ml 0.125% bupivacaine will expand the epidural space.
* In group (B): Bilateral Ultrasound guided Erector spinae group.
* The patient will be in the prone position, after skin sterilization, ESP block will be performed at the level of L3. a curvilinear high-frequency ultrasound transducer will be placed sagittal 3 cm lateral to L3 spinous process where a hyperechoic shadow of the transverse process (TP) and erector spinae will be defined. A 22-gauge spinal needle will be inserted in cranial to caudal direction toward TP in plane to the ultrasound transducer until the needle touches the TP crossing the whole muscles. The location of the needle tip will be confirmed by visible normal saline solution separating erector spinae muscle off the bony shadow of the TP on ultrasound imaging. After confirming the needle site, 30 mL of 0.25% bupivacaine will be injected. The procedure will be repeated following the same steps on the other side.
* Rescue analgesia :

Intra operative :0.5ug /kg of fentanyl as top-up doses at any time if blood pressure and heart rate increased by more than 20% from baseline reading .

Post-operative : Nalbuphine (0.1 mg/kg) will be given if the pain score > 4/10 at the VAS assessment times or when the patient asks for supplementary analgesia due to an emerging pain in between the assessment points.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing Lumbar spine surgery (L1-L5).
* American society of anesthesiologists classification (ASA) I and II.

Exclusion Criteria:

* Patient's refusal.
* Bleeding disorders (platelets count < 150,000; International normalized ratio >1.5; PC< 60%) and coagulopathies.
* Skin lesion, wounds or infection at the injection site.
* Known allergy to local anesthetic drugs.
* Chronic opioid or NSAIDS users.
* Patients with pre-operative opioid consumption

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-05-08 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2023-05-22 (Actual)

PRIMARY OUTCOMES:
time to first analgesia request | 12 hours
  postoperative first rescue analgesia time

SECONDARY OUTCOMES:
cumulative 24 hours opioid consumption | 24 hours
  the total amount of opioid consumed by the patient in the first 24 hours postoperative
presence of any complications | 24 hours
  presence of any complications such as urine retention,vomiting ,respiratory depression
Mean arterial blood pressure | evey 10 minutes intraoperative till end of surgery (up to 2 hours)
  intraoperative mean arterial blood pressure
Heart rate | every 10 minutes intraoperative till end of surgery(up to 2 hours)
  intraoperative heart rate
VAS score | at 15 & 30 mins, then at 2, 6, 12, 24 hours post-operatively
  The visual analog score (VAS) is a validated,subjective measure for acute and chronic pain.scores are recorded by making a handwritten mark on a 10 cm line that represents a continuum between "no pain" and "worst pain"

CONTACTS AND LOCATIONS:
Overall Officials: mohamed F mohamed, ass prof., Study Director — Anesthesia department , Cairo university; Gomaa Z Hussein, professor, Principal Investigator — Anesthesia department , Cairo university
Locations (1):
- Kasr Alainy Hospitals, Giza, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No